CLINICAL TRIAL: NCT03245385
Title: An Open-Label Safety Study to Assess the Multiple-Dose Pharmacokinetics and Potential for Adrenal Suppression Following Topical Treatment With Halobetasol Propionate 0.05% Topical Spray (Sun Pharmaceuticals Industries Limited) in Patients With Moderate to Severe Atopic Dermatitis
Brief Title: Multiple-Dose Pharmacokinetics and Potential for Adrenal Suppression Following Treatment With Halobetasol Spray in Patients With Atopic Dermatitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsors decision
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Collaborators: Novum Pharmaceutical Research Services (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 71542613
Record Dates: First submitted 2017-08-05; First posted 2017-08-10 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Therapeutics; halobetasol

STUDY DESIGN:
Intervention Model Description: Open label, single treatment arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment with topical halobetasol spray 0.05% (Experimental): Patients will instructed o apply halobetasol spray twice daily for 14 days and not to rub over the affected area after application of spray.
  Interventions: Drug: Treatment with Halobetasol propionate 0.05% topical spray

INTERVENTIONS:
Drug: Treatment with Halobetasol propionate 0.05% topical spray — Patients will be treated with topical halobetasol 0.05% spray applied twice daily for 14 days. Patients will be instructed not to rub over the affected area after application of spray. Each patient is expected to receive 28 doses. The maximum amount of test product applied per week will not exceed 50 g

SUMMARY:
This is an open-label, safety study designed to assess the multiple-dose pharmacokinetics and potential for adrenal suppression following topical treatment with halobetasol propionate 0.05% spray applied twice-daily in adult patients with moderate to severe atopic dermatitis. At least 40 eligible patients with atopic dermatitis that satisfy all eligibility criteria will be enrolled into the study

DETAILED DESCRIPTION:
This is an open-label, safety study designed to assess the multiple-dose pharmacokinetics and potential for adrenal suppression following topical treatment with halobetasol propionate 0.05% spray applied twice-daily in adult patients with moderate to severe atopic dermatitis. At least 40 eligible patients with atopic dermatitis that satisfy all eligibility criteria will be enrolled into the study. Patients must be overall in good health and should have a current diagnosis of moderate to severe atopic dermatitis with Investigator Global Assessment (IGA) score of at least 3 or 4. Patients will be stratified by age with:

Cohort 1: At least 20 patients 18 years of age and older with ≥ 25% BSA affected.

Cohort 2: At least 20 patients 12-16 years and 11 months of age with ≥ 25% BSA affected.

Cohort 2 will initiate enrollment once all enrolled patients in Cohort 1 have completed the study and a safety analysis has been reviewed by the Medical Monitor and approved by the Novum Independent Institutional Review Board (NIIRB). Sites will not begin enrollment of patients in Cohort 2 until the site is notified by email that the safety analysis for Cohort 1 has been reviewed and approved. Each cohort will be enrolled based on the availability of patients. Each cohort will be reviewed for the potential of HPA axis suppression. The Medical Monitor or NIIRB may discontinue the study at any time if safety concerns are found. If 6 or more patients in Cohort 1 experience HPA axis suppression, then enrollment for Cohort 1 will be stopped. Cohort 2 will not be initiated if 6 or more patients enrolled in Cohort 1 experience HPA axis suppression or 30% or more of the final enrolled number of patients in Cohort 1 experience HPA axis suppression. If 6 or more patients in Cohort 2 experience HPA axis suppression, then enrollment for Cohort 2 will be stopped. If the study is stopped at any time, patients currently enrolled will be contacted via phone and instructed to discontinue study product immediately. Patients will be instructed to return for their next scheduled visit for cortisol response testing. Sites will follow up with patients and monitor for HPA axis suppression. All patients will be followed until cortisol levels are normal, as defined in study protocol. Patients enrolled in the study will apply the study product twice daily onto the affected skin areas for 14 days (Days 1-14), according to provided instructions. .Patients will be instructed not to rub over the affected area after application of spray. Each patient is expected to receive 28 doses of study product. All patients will attend the clinic for the following 8 scheduled visits. Patients will apply the morning dose of the study product in the clinic at each clinic visit (and evening dose on Day 4) and at home during non-clinic visits. A phone call will be made approximately 14 days after the patient has completed dosing to follow-up on any new adverse events that may have occurred. All patients will have a cortisol response test performed at screening and on Day 17 (at least 48 hours after last dose of study product).

The safety profile of the test product will be evaluated by analysis of reported adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Males or non-pregnant, non-lactating females:

   * Cohort 1: 18 years of age and older
   * Cohort 2: 12-16 years and 11 months of age (Cohort 2 will not begin enrollment until review and approval of safety information from Cohort 1.)
2. If female and of childbearing potential, prepared to abstain from sexual intercourse or use a reliable method of contraception during the study (e.g., condom, IUD, oral, transdermal or injected hormonal contraceptives). Female patients using hormonal contraceptives should have been on the same product/dosing regimen for at least 28 days before baseline and should not change this regimen during the study.
3. Signed informed consent form that meets all criteria of current FDA regulations. For a patient considered to be a minor in the state he/she lives and is enrolled, the parent or legal guardian will be required to sign the consent form and the patient will sign an IRB approved "assent to participate" form. Approved informed consent and assent forms specific to each cohort will be required.
4. Patients with a definite clinical diagnosis of moderate to severe atopic dermatitis with ≥ 25% BSA affected (excluding face, scalp, groin, axillae and other intertriginous areas)
5. Investigator Global Assessment (IGA) score of 3 (Moderate) or 4 (Severe).
6. Patients in Cohort 2 must weigh a minimum of 26 kg.
7. Results from a cortisol response test that are considered normal and show no evidence of any abnormal HPA function or adrenal response. Patients must fulfill all of the following stipulations:

   1. Basal (pre Cortrosyn™ injection) cortisol concentration ≥ 5 mcg/100 mL.
   2. 30-minute post-injection cortisol level is at least 7 mcg/100 mL greater than the basal level (≥ basal value + 7).
   3. Post-stimulation level > 18 mcg/100 mL.

Exclusion Criteria:

1. Females who are pregnant, nursing, planning to become pregnant during the duration of the study, or if of childbearing potential and sexually active and not prepared to use appropriate contraceptive methods to avoid pregnancy.
2. Mild atopic dermatitis.
3. IGA score < 3.
4. Atopic dermatitis with a BSA involvement < 25%.
5. Results from a cortisol response test that show evidence of any abnormal HPA function or adrenal response:

   1. Basal (pre CortrosynTM injection) cortisol concentration < 5 mcg/100 mL.
   2. 30 minute post-injection cortisol level is less than 7 mcg/100 mL greater than the basal level (< basal value + 7).
   3. Post-stimulation level ≤ 18 mcg/100 mL.
6. Recurrent or active cutaneous bacterial or viral infection in any treatment area at baseline (i.e., clinically infected atopic dermatitis).
7. Patient has a history of atopic dermatitis that has been unresponsive to topical corticosteroid therapy.
8. Any condition (i.e., sunburn, psoriasis etc.) that, in the Investigator's opinion, may interfere with the clinical assessments of the signs and symptoms of atopic dermatitis.
9. History of prolonged bleeding or a past diagnosis of bleeding disorders and/or history of blood loss exceeding 450 mL (including blood donations) within 1 month before the study.
10. Patient with poor peripheral venous access.
11. History of mastectomy or lymphatic insufficiency of the upper limb (patient is eligible if blood can be taken from the arm opposite the site of surgery or condition).
12. History of allergy or sensitivity to corticosteroids or history of any drug hypersensitivity or intolerance that, in the opinion of the Investigator, would compromise the safety of the patient or the results of the study.
13. Patient has a significant history or current evidence of chronic infectious disease, system disorder, Netherton's Syndrome, uncontrolled diabetes, organ disorder or insufficiency, immunosuppression (from medical treatment or disease) or other medical condition that, in the Investigator's opinion, would place the study patient at undue risk by participation in the study or as an unsuitable candidate for pharmacokinetic blood sampling.
14. Patient is currently receiving or has received any radiation therapy or anti-neoplastic agents within 3 months before baseline.
15. Use within 4 weeks before baseline of 1) oral or intravenous corticosteroids, 2) UVA/UVB therapy, 3) PUVA (psoralen plus ultraviolet A therapy, 4) topical tacrolimus, 5) topical pimecrolimus, 6) systemic retinoids or 7) any other systemic atopic dermatitis treatment.
16. Known history of hypothalamic-pituitary-adrenal axis impairment or any other disturbance of the adrenal function (e.g., Cushing or Addison disease).
17. Use of tanning booths or nonprescription UV light source within 2 weeks before baseline.
18. Use within 8 weeks before baseline of 1) immunomodulators or immunosuppressive therapies or 2) interferon.
19. Use within 14 days before baseline of 1) systemic antibiotics, 2) calcipotriene or other Vitamin D preparations, or 3) topical retinoids.
20. Patients who have used topical treatments, prescription or over the counter, including:

    1. Any topical atopic dermatitis therapeutic agents of any kind within the 2 weeks before baseline.
    2. Any topical corticosteroids within the 2 weeks before baseline.
    3. Any antibacterial, medicated and/or astringent washes, soaps, pads or moisturizers within 3 days before baseline.
    4. High strength (20% or above) alpha-hydroxy acid or any kind of peel or other procedures (e.g., laser hair removal) within 30 days before baseline.
    5. Any topical products (i.e., sunscreens, lotions, creams), except for bland emollient (moisturizer) within 24 hour before baseline.
    6. Topical antibiotics in the treatment area within 7 days before baseline.
21. Patient has been treated within 6 months before baseline with any biological therapies for atopic dermatitis.
22. Inability to understand the protocol requirements, instructions, and study-related restrictions, the nature, scope, and possible consequences of the clinical study.
23. Unlikely to comply with the protocol requirements, instructions, and study-related restrictions, such as uncooperative attitude, inability to return for follow-up visits, and improbability of completing the clinical study.
24. Receipt of any drug as part of a research study within 30 days before baseline.
25. The patient is a member of the investigational study staff or a member of the family of the investigational study staff.
26. Previous participation in this study.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2018-02-05 (Actual); Study Completion 2018-02-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the IGA score at Days 4, 5, 7 and 14. | 14 days
  Patients will be considered to have shown improvement in disease severity if the IGA score decreases by at least one unit from the baseline score, and will be considered a treatment success if the IGA score is either 0 (clear) or 1 (almost clear).

SECONDARY OUTCOMES:
Hypothalamic Pituitary Adrenal (HPA) Axis suppression | 14 days
  Hypothalamic Pituitary Adrenal (HPA) Axis Response to Cosyntropin demonstrating the absence or presence, defined by 30 minute post- CortrosynTM injection level cortisol level of ≤18 mcg/100 mL, at the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Rajinder K Jalali, MD, Study Director — Sun Pharmaceutical Industries Limited
Locations (13):
- United States (13):
  - Providence Clinical Research, North Hollywood, California
  - Havana Research Institute, Pasadena, California
  - Vital Pharma Research, Hialeah, Florida
  - Solutions Through Advanced Research, Jacksonville, Florida
  - Integrity Research Center, Miami, Florida
  - Millennium Clinical Research, INC, Miami, Florida
  - Regenerate Clinical Trials, LLC, Miami, Florida
  - Life Medical Center and Research, INC, Miami, Florida
  - Vista Health Research, Miami, Florida
  - Elias Research, Troy, Michigan
  - Montana Medical Research/Elias Research Assoc., Missoula, Montana
  - L&C Professional Medical Research Institute, Hazleton, Pennsylvania
  - Sun Research Institute, San Antonio, Texas